CLINICAL TRIAL: NCT05569759
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2a Study With Open-label Extension to Evaluate the Safety and Efficacy of Zetomipzomib (KZR-616) in Patients With Autoimmune Hepatitis
Brief Title: A Study of Zetomipzomib (KZR-616) in Patients With Autoimmune Hepatitis (PORTOLA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kezar Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KZR-616-208
Record Dates: First submitted 2022-09-29; First posted 2022-10-06 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Autoimmune Hepatitis
Keywords: immunoproteasome inhibition; selective proteasome inhibition; disease flare; liver enzymes; ALT (alanine aminotransferase); AST (aspartate aminotransferase); glucocorticoids; steroids
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — KZR-616; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- zetomipzomib + standard-of-care (glucocorticoids) (Experimental): Initial 30 mg dose of zetomipzomib, followed by weekly 60 mg doses of zetomipzomib, for the remaining 23 weeks of the treatment period.
  Interventions: Drug: zetomipzomib
- placebo + standard-of-care (glucocorticoids) (Placebo Comparator): Initial 30 mg dose of placebo (sterile water for injection), followed by weekly 60 mg doses of placebo, for the remaining 23 weeks of the treatment period.
  Interventions: Drug: placebo
- zetomipzomib + standard-of care (glucocorticoids) open-label extension period (Experimental): Initial 30 mg dose of zetomipzomib at the open-label extension (OLE) Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib, for up to a total of 24 additional weeks of treatment.
  Interventions: Drug: zetomipzomib in open-label extension

INTERVENTIONS:
Drug: zetomipzomib — Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
  Other Names: KZR-616
  Arms: zetomipzomib + standard-of-care (glucocorticoids)
Drug: placebo — Subcutaneous injection of placebo
  Other Names: sterile water for injection
  Arms: placebo + standard-of-care (glucocorticoids)
Drug: zetomipzomib in open-label extension — Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
  Other Names: KZR-616
  Arms: zetomipzomib + standard-of care (glucocorticoids) open-label extension period

SUMMARY:
This was a Phase 2a, multi-center, placebo-controlled study in which patients with autoimmune hepatitis received zetomipzomib or placebo in addition to standard-of-care for 24 weeks; an optional open-label extension period allowed participants to receive zetomipzomib (KZR-616) for an additional 24 weeks of treatment.

DETAILED DESCRIPTION:
This was a Phase 2a, multi-center, randomized, double-blind, placebo-controlled study with an open-label extension to evaluate safety, tolerability, and efficacy of zetomipzomib in patients with autoimmune hepatitis (AIH) who have not benefited from standard-of-care treatment, had an incomplete response to ≥3 months of standard-of-care treatment, or had a disease flare after standard of care.

Zetomipzomib or placebo were administered weekly for a 24-week treatment period in addition to standard-of-care (glucocorticoids), followed by a 4-week off-treatment safety follow-up period. Zetomipzomib and placebo was administered subcutaneously (SC) once weekly.

At the end of the 24-week treatment period, eligible participants from both the zetomipzomib- and placebo-treated arms who completed the double-blind treatment period could enroll in the open-label extension period to receive up to an additional 24 weeks of treatment with zetomipzomib.

ELIGIBILITY:
Key Inclusion Criteria for the Double-blind Treatment Period:

* Must be aged ≥18 years.

  * Must have a clinical diagnosis of AIH and signs of active disease despite standard-of-care therapy for ≥3 months or disease flare after experiencing complete remission induced by standard-of-care treatment, including:

    * Screening ALT values that are 1.25 to 10 times the upper limit of the normal range (ULN)
    * Liver biopsy results with Ishak score (modified HAI) ≥5/18 indicating active AIH, from a biopsy performed at Screening, or within 6 months prior to Screening
    * Mild or no hepatic impairment (Child Pugh category A)
  * Must be willing to use and taper glucocorticoid therapy.
  * Must be willing to use effective contraception.

Key Exclusion Criteria for the Double-blind Treatment Period:

* Have a concomitant diagnosis of primary biliary sclerosis, primary sclerosing cholangitis, IgG 4 related cholangitis, drug related AIH (at Screening) or a history of drug-related AIH.
* Have clinical evidence of significant unstable or uncontrolled diseases other than the disease under study.
* Are receiving oral or injectable immunomodulating treatment for any other autoimmune disease prior to enrollment in the study. Patients who have been using such treatments must follow the specified washout periods.
* Have an active infection (eg, acute hepatitis E, cytomegalovirus, or Epstein-Barr virus) requiring systemic therapy with antibiotic, antiviral, or antifungal treatment, or has had any febrile illness within 7 days prior to Day -1.
* Have a history of thyroiditis, celiac disease, or other autoimmune disorder known to be associated with transaminitis.
* Have liver cirrhosis with significant impairment of liver function (Child Pugh category B or C) or have decompensated cirrhosis.
* Patients with histology confirmed coincident non-alcoholic steatohepatitis.

Key Inclusion Criteria for the Open-label Extension Period:

* Same as Double-blind Treatment Period inclusion criteria, except the following modifications:

  * ALT value can be normal or, if elevated, in the range of 1.25 to 10 times the upper limit of normal
* Must have completed the Double-blind Period study visits through Week 24, including all Week 24 Visit assessments.
* Must be willing to maintain glucocorticoid therapy or continue to taper glucocorticoid therapy.

Key Exclusion Criteria for the Open-label Extension Period:

• Same as Double-blind Treatment Period except no need to re-test for HIV, HBV, HCV, and TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Lammert, MD, Principal Investigator — Indiana University; Ethan Weinberg, MD, Principal Investigator — University of Pennsylvania
Locations (24):
- United States (24):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Keck School of Medicine of USC, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford Medicine, Redwood City, California
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health Center for Liver Disease and Transplantation, Manhasset, New York
  - New York University Langone Health/Grossman School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Corporate website — https://www.kezarlifesciences.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The randomization stratification factor for the study was use of glucocorticoids at Screening (ie, glucocorticoid use, no glucocorticoid use at Screening).
Groups:
- Zetomipzomib + Standard-of-care (Glucocorticoids): Participants received an initial 30 mg dose of zetomipzomib, followed by weekly 60 mg doses of zetomipzomib, for the remaining 23 weeks of the treatment period in addition to standard of care.
  Participants who completed the double blind treatment period could elect to continue in the open-label extension (OLE) period of the study. Participants who enrolled in the OLE period received an initial 30 mg dose of zetomipzomib at the open-label extension (OLE) Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib in addition to standard of care, for up to a total of 24 additional weeks of treatment.
  zetomipzomib: Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
- Placebo + Standard-of-care (Glucocorticoids): Participants received an initial 30 mg dose of placebo (sterile water for injection), followed by weekly 60 mg doses of placebo, for the remaining 23 weeks of the treatment period in addition to standard of care.
  placebo: Subcutaneous injection of placebo
  Participants who completed the double blind treatment period could elect to continue in the open-label extension (OLE) period of the study. Participants who enrolled in the OLE period received an initial 30 mg dose of zetomipzomib at the open-label extension (OLE) Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib in addition to standard of care, for up to a total of 24 additional weeks of treatment.
Period: Double Blind Treatment Period
Arm/Group | Zetomipzomib + Standard-of-care (Glucocorticoids) | Placebo + Standard-of-care (Glucocorticoids)
Started | 16 | 8
Completed | 13 | 7
Not Completed | 3 | 1
Period: Optional Open-Label Extension
Arm/Group | Zetomipzomib + Standard-of-care (Glucocorticoids) | Placebo + Standard-of-care (Glucocorticoids)
Started | 9 | 5
Completed | 4 | 3
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are presented for the Full Analysis Set (N=23), all randomized patients who received at least 1 dose of IMP in this study and have Baseline and at least one post-treatment value for all the following measures: ALT, AST, and IgG. One participant was randomized to the placebo group but never dosed and is therefore not included in the Full Analysis Set or the Safety Analysis Set but is included in the Intent to Treat Analysis Set.
Groups:
- Zetomipzomib + Standard-of-care (Glucocorticoids): Participants received an initial 30 mg dose of zetomipzomib, followed by weekly 60 mg doses of zetomipzomib, for the remaining 23 weeks of the double-blind treatment period in addition to standard of care.
  Participants who completed the double-blind treatment period could elect to continue in the open-label extension (OLE) period of the study. Participants who enrolled in the OLE period received an initial 30 mg dose of zetomipzomib at the OLE Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib in addition to standard of care, for up to a total of 24 additional weeks of treatment.
  zetomipzomib: Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
- Placebo + Standard-of-care (Glucocorticoids): Participants received an initial 30 mg dose of placebo (sterile water for injection), followed by weekly 60 mg doses of placebo, for the remaining 23 weeks of the double-blind treatment period in addition to standard of care.
  placebo: Subcutaneous injection of placebo
  Participants who completed the double-blind treatment period could elect to continue in the open-label extension (OLE) period of the study. Participants who enrolled in the OLE period received an initial 30 mg dose of zetomipzomib at the OLE Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib in addition to standard of care, for up to a total of 24 additional weeks of treatment.
- Total: Total of all reporting groups
Arm/Group | Zetomipzomib + Standard-of-care (Glucocorticoids) | Placebo + Standard-of-care (Glucocorticoids) | Total
Number analyzed (Participants) | 16 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (15.6) | 48.9 (19.7) | 52.7 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 8 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 14 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  Native Hawaiian | 0 | 0 | 0
  White | 13 | 6 | 19
  Asian Indian | 0 | 0 | 0
  Chinese | 0 | 0 | 0
  Filipino | 0 | 0 | 0
  Japanese | 0 | 0 | 0
  Korean | 0 | 0 | 0
  Vietnamese | 0 | 0 | 0
  Other Asian | 0 | 0 | 0
  Guamanian or Chamorro | 0 | 0 | 0
  Samoan | 0 | 0 | 0
  Other Pacific Islander | 0 | 0 | 0
  Other | 2 | 0 | 2
  Multi-Racial | 0 | 0 | 0
Baseline ALT [Mean (Standard Deviation); unit: U/L] | 106.7 (49.0) | 143.4 (75.2) | 117.9 (59.0)
Baseline AST [Mean (Standard Deviation); unit: U/L] | 79.5 (50.4) | 107.0 (40.6) | 87.8 (48.4)
Baseline IgG [Mean (Standard Deviation); unit: mg/dL] | 1865.3 (842.5) | 1985.1 (579.2) | 1901.7 (760.7)
Baseline IgG (Abnormal at Baseline) [Mean (Standard Deviation); unit: mg/dL] — Population: This is the subset of participants with abnormal baseline IgG values.
  mg/dL
    number analyzed (Participants) | 9 | 5 | 14
    (all) | 2396.7 (751.8) | 2213.0 (514.5) | 2331.1 (661.5)
Duration of AIH [Mean (Standard Deviation); unit: years] | 5.5 (5.9) | 8.3 (7.6) | 6.3 (6.4)
Glucocorticoid Dose at Baseline [Mean (Standard Deviation); unit: mg/day] | 21.3 (3.4) | 20.0 (0.0) | 20.9 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Achieved Complete Biochemical Response
Description: The number of patients who achieve complete biochemical response (CR), defined as normal ALT, AST, and IgG values (if IgG level is elevated at Baseline) with glucocorticoid dose not higher than starting dose (at Baseline), by Week 24 of the Double-Blind Treatment Period. Analyses were also conducted at Week 12, Week 16, and Week 20.
Time Frame: Week 12, Week 16, Week 20, and Week 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids): Participants received an initial 30 mg dose of zetomipzomib, followed by weekly 60 mg doses of zetomipzomib, for the remaining 23 weeks of the treatment period in addition to standard of care during the double-blind treatment period.
  zetomipzomib: Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
- Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids): Participants received an initial 30 mg dose of placebo (sterile water for injection), followed by weekly 60 mg doses of placebo, for the remaining 23 weeks of the treatment period in addition to standard of care during the double-blind treatment period.
  placebo: Subcutaneous injection of placebo
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
Participants
  Week 12 | 6 | 3
  Week 16 | 7 | 3
  Week 20 | 8 | 3
  Week 24 | 8 | 3

2. Primary Outcome: The Safety and Tolerability of Zetomipzomib
Description: Proportion of participants who experience AEs (adverse events) and SAEs (serious adverse events) during the double-blind treatment period (DBTP) and the open-label extension (OLE).
Time Frame: Baseline through end of study visit (DBTP, Week 28 and OLE, Up to Week 24)
Population: The Safety Set (N=23) includes all participants who received at least one dose of IMP and were analyzed as randomized to treatment.
Measure: Number; unit: participants
Groups:
- Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids): Participants received an initial 30 mg dose of zetomipzomib, followed by weekly 60 mg doses of zetomipzomib, for the remaining 23 weeks of the double-blind treatment period in addition to standard of care.
  zetomipzomib in the double-blind treatment period: Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
- Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids): Participants received an initial 30 mg dose of placebo (sterile water for injection), followed by weekly 60 mg doses of placebo, for the remaining 23 weeks of the double-blind treatment period in addition to standard of care.
  placebo in the double-blind treatment period: Subcutaneous injection of placebo
- Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Zetomipzomib in DBTP): Participants, who received zetomipzomib in the double-blind treatment period (DBTP) and enrolled in the open-label extension period, received an initial 30 mg dose of zetomipzomib at the open-label extension (OLE) Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib, for up to a total of 24 additional weeks of treatment in addition to standard of care.
  zetomipzomib in open-label extension who received zetomipzomib during the double-blind treatment period: Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
- Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Placebo in DBTP): Participants, who received placebo in the double-blind treatment period (DBTP) and enrolled in the open-label extension period, received an initial 30 mg dose of zetomipzomib at the open-label extension (OLE) Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib, for up to a total of 24 additional weeks of treatment in addition to standard of care.
  zetomipzomib in open-label extension who received placebo during the double-blind treatment period: Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Zetomipzomib in DBTP) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Placebo in DBTP)
Number analyzed (Participants) | 16 | 7 | 9 | 5
participants
  Serious adverse events | 2 | 1 | 0 | 0
  Adverse events | 16 | 7 | 9 | 5

3. Primary Outcome: Proportion of Participants Experiencing a Disease Flare Among the Participants Who Achieved a CR During the Double-blind Treatment Period
Description: Proportion of participants experiencing a disease flare among the participants who achieved a complete biochemical response (CR) during the double-blind treatment period.
Time Frame: Start of open-label extension (OLE) period through End of Study (EOS) up to OLE Week 25
Population: Participants who enrolled in the optional open-label extension following their completion of the double-blind treatment period of the study and achieved a complete response during the double-blind treatment period.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Zetomipzomib in DBTP) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Placebo in DBTP)
Number analyzed (Participants) | 5 | 2
participants | 0 [0.0 to 52.2] | 0 [0.0 to 84.2]

4. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: Changes from baseline in alanine aminotransferase (ALT) during the double-blind treatment period.
Time Frame: Weeks 12, 16, 20, and 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
U/L
  Week 12 | -49.8 (67.1) | -47.3 (116.5)
  Week 16 | -46.4 (70.4) | -65.8 (81.7)
  Week 20 | -29.4 (100.8) | -33.3 (113.4)
  Week 24 | -22.8 (103.5) | -80.6 (58.0)

5. Secondary Outcome: Partial Response
Description: Proportion of participants who achieved a partial response (PR) during the double-blind treatment period of the study.
Time Frame: Weeks 12, 16, 20, and 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
Participants
  Week 12 | 4 | 2
  Week 16 | 1 | 0
  Week 20 | 1 | 0
  Week 24 | 2 | 1

6. Secondary Outcome: Time to Complete Response
Description: Time to complete response (CR), defined as the duration from first dose of study drug (zetomipzomib or placebo) to first CR, during the double-blind treatment period was measured using the Kaplan-Meier method. Due to the small sample size, not enough events of participants achieving CR were observed to provide Kaplan-Meier estimates for the 25th percentile, median, and 75th percentile time to CR.
Time Frame: Baseline through Week 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
weeks | NA [8.14 to NA] — Not evaluable due to the small number of participants who achieved complete response as participants who did not achieve a CR were considered non-responders and were censored from analysis. | NA [4.14 to NA] — Not evaluable due to the small number of participants who achieved complete response as participants who did not achieve a CR were considered non-responders and were censored from analysis.

7. Secondary Outcome: Disease Flare After CR
Description: Proportion of participants who experienced a disease flare after complete response (CR) during the double-blind treatment period.
Time Frame: Week 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
Participants | 0 | 0

8. Secondary Outcome: Treatment Failures
Description: Proportion of participants who were considered treatment failures, defined as ALT or AST level worsened ≥2 times that of the Baseline value that is sustained for ≥1 week as verified via repeat laboratory assessments, despite compliance with standard of care (ie, with regard to inclusion criteria) or protocol-defined therapy or a glucocorticoid dose is increased above the Baseline dose, it may be considered a treatment failure unless attributed to an adverse event not relating to AIH, during the double-blind treatment period.
Time Frame: Week 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
Participants | 2 | 1

9. Secondary Outcome: Complete Response With Glucocorticoid Taper to ≤10 mg
Description: Percentage of participants who achieved complete response with successful glucocorticoid taper to ≤10 mg by Week 24 of the double-blind treatment period.
Time Frame: Weeks 12, 16, 20, and 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
percent of participants
  By Week 12 | 18.8 [4.0 to 45.6] | 25.0 [3.2 to 65.1]
  By Week 16 | 37.5 [15.2 to 64.6] | 25.0 [3.2 to 65.1]
  By Week 20 | 43.8 [19.8 to 70.1] | 25.0 [3.2 to 65.1]
  By Week 24 | 43.8 [19.8 to 70.1] | 25.0 [3.2 to 65.1]

10. Secondary Outcome: Complete Response With Glucocorticoid Taper to ≤5 mg
Description: Percentage of participants who achieved complete response and glucocorticoid taper to ≤5 mg by Week 24 of the double-blind treatment period.
Time Frame: Weeks 12, 16, 20, and 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
percent of participants
  By Week 12 | 12.5 [1.6 to 38.3] | 0 [0 to 36.9]
  Be Week 16 | 25.0 [7.3 to 52.4] | 12.5 [0.3 to 52.7]
  By Week 20 | 37.5 [15.2 to 64.6] | 12.5 [0.3 to 52.7]
  By Week 24 | 37.5 [15.2 to 64.6] | 12.5 [0.3 to 52.7]

11. Secondary Outcome: Complete Response With Glucocorticoid Taper to 0 mg
Description: Percentage of participants who achieved complete response with glucocorticoid taper to 0 mg by Week 24 of the double-blind treatment period.
Time Frame: Weeks 12, 16, 20, and 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
percent of participants
  By Week 12 | 6.3 [0.2 to 30.2] | 0 [0.0 to 36.9]
  By Week 16 | 6.3 [0.2 to 30.2] | 0 [0.0 to 36.9]
  By Week 20 | 12.5 [1.6 to 38.3] | 0 [0.0 to 36.9]
  By Week 24 | 25.0 [7.3 to 52.4] | 0 [0.0 to 36.9]

12. Secondary Outcome: Partial Response With Glucocorticoid Taper to ≤10 mg
Description: Percentage of participants who achieved partial response with successful glucocorticoid taper to ≤10 mg by Week 24 of the double-blind treatment period.
Time Frame: Week 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
percent of participants | 31.3 [11.0 to 58.7] | 25.0 [3.2 to 65.1]

13. Secondary Outcome: Partial Response With Glucocorticoid Taper to ≤5 mg
Description: Percentage of participants who achieved partial response and glucocorticoid taper to ≤5 mg by Week 24 of the double-blind treatment period.
Time Frame: Week 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
percent of participants | 12.5 [1.6 to 38.3] | 12.5 [0.3 to 52.7]

14. Secondary Outcome: Partial Response With Glucocorticoid Taper to 0 mg
Description: Percentage of participants who achieved partial response with glucocorticoid taper to 0 mg by Week 24 of the double-blind treatment period.
Time Frame: Week 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
percent of participants | 12.5 [1.6 to 38.3] | 0 [0.0 to 36.9]

15. Other Pre Specified Outcome: Change From Baseline in Glucocorticoid Dose
Description: Mean change from Baseline in glucocorticoid dose for participants during the double-blind treatment period at Weeks 12, 16, 20 and 24
Time Frame: Weeks 12, 16, 20, and 24
Population: The Intent to Treat (ITT) Set included all randomized participants (N=24).
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 16 | 8
mg/day
  Week 12: number analyzed (Participants) | 15 | 7
  Week 12 | -6.2 (9.44) | -3.2 (11.70)
  Week 16: number analyzed (Participants) | 15 | 7
  Week 16 | -8.3 (10.59) | -3.0 (13.83)
  Week 20: number analyzed (Participants) | 14 | 6
  Week 20 | -10.0 (11.35) | -7.2 (10.30)
  Week 24: number analyzed (Participants) | 13 | 7
  Week 24 | -12.5 (9.79) | -4.7 (11.43)

16. Post Hoc Outcome: Complete Response With Glucocorticoid Taper to ≤10 mg (Subset of Participants on Steroids at Screening)
Description: For the subset of the intent to treat population who were on glucocorticoid steroids at Screening, the percentage of participants who achieved complete response with successful glucocorticoid taper to ≤10 mg by Week 24 of the double-blind treatment period is presented.
Time Frame: Weeks 12, 16, 20, and 24
Population: The subset of participants in the intent to treat population who were on glucocorticoids at Screening.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 14 | 7
percent of participants
  By Week 12 | 21.4 [4.7 to 50.8] | 14.3 [0.4 to 57.9]
  By Week 16 | 42.9 [17.7 to 71.1] | 14.3 [0.4 to 57.9]
  By Week 20 | 50.0 [23.0 to 77.0] | 14.3 [0.4 to 57.9]
  By Week 24 | 50.0 [23.0 to 77.0] | 14.3 [0.4 to 57.9]

17. Post Hoc Outcome: Complete Response With Glucocorticoid Taper to ≤5 mg (Subset of Participants on Steroids at Screening)
Description: For the subset of the intent to treat population who were on glucocorticoid steroids at Screening, the percentage of participants who achieved complete response with successful glucocorticoid taper to ≤5 mg by Week 24 of the double-blind treatment period is presented.
Time Frame: Weeks 12, 16, 20, and 24
Population: The subset of participants in the intent to treat population who were on glucocorticoids at Screening. Of note, one participant met the SAP definition of CR with glucocorticoid taper to 0 mg at Week 4 with normalized ALT, AST, and IgG while taking no glucocorticoid steroids and is included in this dataset. After further review of the data, notes in the database stated the reason for the participant taking no glucocorticoids for 7 days was due to the glucocorticoid medication unavailability.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 14 | 7
percent of participants
  By Week 12 | 14.3 [1.8 to 42.8] | 0 [0.0 to 41.0]
  By Week 16 | 28.6 [8.4 to 58.1] | 0 [0.0 to 41.0]
  By Week 20 | 42.9 [17.7 to 71.1] | 0 [0.0 to 41.0]
  By Week 24 | 42.9 [17.7 to 71.1] | 0 [0.0 to 41.0]

18. Post Hoc Outcome: Complete Response With Glucocorticoid Taper to 0 mg (Subset of Participants on Steroids at Screening)
Description: For the subset of the intent to treat population who were on glucocorticoid steroids at Screening, the percentage of participants who achieved complete response with successful glucocorticoid taper to 0 mg by Week 24 of the double-blind treatment period is presented.
Time Frame: Weeks 12, 16, 20, and 24
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 14 | 7
percent of participants
  By Week 12 | 7.1 [0.2 to 33.9] | 0 [0.0 to 41.0]
  By Week 16 | 7.1 [0.2 to 33.9] | 0 [0.0 to 41.0]
  By Week 20 | 14.3 [1.8 to 42.8] | 0 [0.0 to 41.0]
  By Week 24 | 28.6 [8.4 to 58.1] | 0 [0.0 to 41.0]

19. Post Hoc Outcome: Complete Response (Subset of Participants on Steroids at Screening)
Description: For the subset of the intent to treat population who were on glucocorticoid steroids at Screening, the percentage of participants who achieved complete response by Week 24 of the double-blind treatment period is presented.
Time Frame: Weeks 12, 16, 20, and 24
Population: The subset of participants in the intent to treat population who were on glucocorticoids at Screening.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids)
Number analyzed (Participants) | 14 | 7
percent of participants
  Week 12 | 42.9 [17.7 to 71.1] | 28.6 [3.7 to 71.0]
  Week 16 | 50.0 [23.0 to 77.0] | 28.6 [3.7 to 71.0]
  Week 20 | 57.1 [28.9 to 82.3] | 28.6 [3.7 to 71.0]
  Week 24 | 57.1 [28.9 to 82.3] | 28.6 [3.7 to 71.0]

ADVERSE EVENTS:
Time Frame: 28 weeks during the double-blind treatment period and up to an additional 28 weeks for participants enrolled in the optional open label extension period
Groups:
- Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Zetomipzomib in DBTP): Participants, who received zetomipzomib in the double-blind treatment period (DBTP) and enrolled in the open-label extension period, received an initial 30 mg dose of zetomipzomib at the open-label extension (OLE) Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib, for up to a total of 24 additional weeks of treatment in addition to standard of care.
  zetomipzomib in OLE who received zetomipzomib during the DBTP: Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
- Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Placebo in DBTP): Participants, who received placebo in the double-blind treatment period (DBTP) and enrolled in the open-label extension period, received an initial 30 mg dose of zetomipzomib at the open-label extension (OLE) Week 1 visit, followed by weekly doses of 60 mg of zetomipzomib, for up to a total of 24 additional weeks of treatment in addition to standard of care.
  zetomipzomib in OLE who received placebo during the DBTP: Subcutaneous injection of zetomipzomib with a target dose of 60 mg weekly
Arm/Group | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Zetomipzomib in DBTP) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Placebo in DBTP)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/7 | 0/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/7 | 0/9 | 0/5
Other Adverse Events (participants affected / at risk) | 16/16 | 7/7 | 9/9 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) (N=16) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids) (N=7) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Zetomipzomib in DBTP) (N=9) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Placebo in DBTP) (N=5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind Treatment Period: Zetomipzomib + Standard-of-care (Glucocorticoids) (N=16) | Double-blind Treatment Period: Placebo + Standard-of-care (Glucocorticoids) (N=7) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Zetomipzomib in DBTP) (N=9) | Open-label Extension: Zetomipzomib + standard-of Care (Glucocorticoids) (Placebo in DBTP) (N=5)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (14) | 0 (0) | 2 (5) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (5) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (23) | 2 (7) | 4 (10) | 3 (12)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (7) | 1 (1) | 2 (3) | 0 (0)
Application site purpura (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders and administration site conditions) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders and administration site conditions) | 9 (34) | 2 (12) | 6 (22) | 4 (21)
Cyst (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders and administration site conditions) | 6 (28) | 3 (3) | 4 (6) | 2 (10)
Influenza like illness (General disorders and administration site conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders and administration site conditions) | 7 (19) | 4 (8) | 2 (2) | 1 (1)
Injection site discolouration (General disorders and administration site conditions) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Injection site discomfort (General disorders and administration site conditions) | 2 (4) | 1 (6) | 0 (0) | 1 (9)
Injection site erythema (General disorders and administration site conditions) | 12 (76) | 2 (3) | 3 (14) | 3 (31)
Injection site exfoliation (General disorders and administration site conditions) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site hypoaesthesia (General disorders and administration site conditions) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders and administration site conditions) | 5 (40) | 0 (0) | 1 (2) | 4 (22)
Injection site inflammation (General disorders and administration site conditions) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders and administration site conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site nodule (General disorders and administration site conditions) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Injection site pain (General disorders and administration site conditions) | 10 (50) | 1 (2) | 3 (8) | 3 (4)
Injection site papule (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site paraesthesia (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders and administration site conditions) | 7 (54) | 0 (0) | 3 (11) | 2 (11)
Injection site rash (General disorders and administration site conditions) | 5 (9) | 0 (0) | 1 (1) | 2 (2)
Injection site swelling (General disorders and administration site conditions) | 5 (10) | 0 (0) | 2 (4) | 0 (0)
Injection site urticaria (General disorders and administration site conditions) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site vesicles (General disorders and administration site conditions) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Injection site warmth (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Malaise (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders and administration site conditions) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders and administration site conditions) | 6 (13) | 3 (3) | 5 (5) | 1 (2)
Peripheral swelling (General disorders and administration site conditions) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders and administration site conditions) | 8 (23) | 2 (2) | 4 (5) | 2 (9)
Swelling face (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders and administration site conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders and administration site conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site bruising (General disorders and administration site conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ocular icterus (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 0 (0) | 1 (2)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural pruritus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (6) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cranial nerve neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain fog (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (42) | 4 (9) | 4 (10) | 3 (8)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Listless (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0) | 4 (9) | 1 (12)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (2) | 1 (1) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (7) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Peripheral vascular haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of this study include its small sample size, unpowered design, and a predominantly white study population, which may limit generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT05569759/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT05569759/SAP_001.pdf